CLINICAL TRIAL: NCT06304441
Title: A Clinical Trial of Intra-pemetrexed Plus Third-generation Small Molecule TKI Drugs (e.g. 'Osimertinib') Versus Third-generation Small Molecule TKI Drugs Alone for Leptomeningeal Metastasis From Epidermal Growth Factor Receptor Mutation-Positive Non-Small-cell Lung Cancer
Brief Title: Intra-pemetrexed Plus Third-generation Small Molecule TKI Drugs (e.g. 'Osimertinib') Versus Third-generation Small Molecule TKI Drugs Alone for Leptomeningeal Metastasis From Epidermal Growth Factor Receptor Mutation-Positive Non-Small-cell Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Zhenyu Pan, Professor, Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPVO
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Leptomeningeal Metastasis
Keywords: Leptomeningeal metastasis; Intrathecal chemotherapy; Pemetrexed; Third-generation small molecule TKI drugs; Osimertinib; Epidermal growth factor receptor mutation
MeSH Terms: conditions — Meningeal Carcinomatosis | interventions — osimertinib; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Intra-pemetrexed plus third-generation small molecule TKI drugs (e.g. 'osimertinib')
  Interventions: Drug: Osimertinib; Drug: Pemetrexed
- Group B (Active Comparator): Third-generation small molecule TKI drugs (e.g. 'osimertinib') alone
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — Double-dose of TKI (e.g. 'osimertinib' 160 mg) was administered orally once daily until disease progression or unmanageable drug-related toxicity.
Drug: Pemetrexed — Pemetrexed 15 mg was administered with dexamethasone 5 mg via intraventricular or via lumbar puncture. First, induction intrathecal chemotherapy, twice per week for 2 weeks; then consolidation intrathecal chemotherapy, once per week for 4 weeks; and maintenance intrathecal chemotherapy, once per month until disease progression or unmanageable drug-related toxicity.
  Arms: Group A

SUMMARY:
Intrathecal chemotherapy is one of the mainstay treatment options for leptomeningeal metastases. Pemetrexed is one of the first-line chemotherapeutic agents for non-squamous non-small cell lung cancer (NSCLC). Since 2017, intrathecal pemetrexed has shown good efficacy for patients with leptomeningeal metastases from NSCLC. It has been recommended as the preferred drug for intrathecal chemotherapy by the Chinese Society of Clinical Oncology (CSCO) guidelines. Tyrosine kinase inhibitors (TKIs) play a promising role in the treatment of non-small cell lung cancer patients with epidermal growth factor receptor (EGFR) mutations. Due to its small molecule properties, it can effectively penetrate the central nervous system barrier and deliver an effective antitumor effect. An international multi-center clinical study published in 2019 confirmed that double-dose of osimertinib showed significant improvement in leptomeningeal metastases from NSCLC with EGFR exon 19 deletion or exon 21 L858R/T790M mutation. It makes TKIs the mainstay of treatment for patients with EGFR-mutant NSCLC with leptomeningeal metastases. However, whether third-generation small molecule TKI drugs (e.g. 'osimertinib') combined with intrathecal pemetrexed could benefit patients with LM from EGFR- mutant NSCLC remains undetermined.

DETAILED DESCRIPTION:
The aim of this Study is to compare the effects of intra-pemetrexed Plus third-generation small molecule TKI drugs (e.g. 'osimertinib') versus third-generation small molecule TKI drugs alone in leptomeningeal metastasis from EGFR mutation positive NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged between 18 and 75 years.
2. Histologically or cytologically confirmed diagnosis of NSCLC with single activating EGFR mutations (L858R or Exon19Del).
3. Confirmed diagnosis of leptomeningeal metastasis according to ESMO/EANO guidelines.
4. Normal liver and kidney function; WBC≥4000/mm3, Plt≥100000/mm3.
5. No history of severe nervous system disease.
6. No severe dyscrasia.

Exclusion Criteria:

1. Any evidence of nervous system failure, including severe encephalopathy, grade 3 or 4 leukoencephalopathy on imaging, and Glasgow Coma Score less than 11.
2. Any evidence of extensive and lethal progressive systemic diseases without effective treatment.
3. Patients with poor compliance or other reasons that were unsuitable for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Clinical response rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months.
  The response assessment in neuro-oncology criteria (RANO) proposal for response criteria of leptomeningeal metastasis was used to assess the clinical response in this study.

SECONDARY OUTCOMES:
Overall survival | From the enrollment of this study until date of death from any cause, whichever came first, or the last follow-up (at least 7 months).
  Survival time was recorded since the date of patient enrollment. All patients were followed up until death or the end of the study.
Incidence of treatment-related adverse events | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months.
  The incidence of treatment-related adverse events were measured for determining tolerability and safety. Adverse events (AEs) are evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE, version 4.03).
  Events of grade 3-5 are defined as moderate and severe adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third People's Hospital of Huizhou (Huizhou Hospital of Guangzhou Medical University), Huizhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Starting 6 months after publication.
Access Criteria: Individual participant data will be public accessable via contacting with principal investigator by email within 6 months after the trial complete.

REFERENCES:
- [Background] Pan Z, Yang G, He H, Cui J, Li W, Yuan T, Chen K, Jiang T, Gao P, Sun Y, Cong X, Li Z, Wang Y, Pang X, Song Y, Zhao G. Intrathecal pemetrexed combined with involved-field radiotherapy as a first-line intra-CSF therapy for leptomeningeal metastases from solid tumors: a phase I/II study. Ther Adv Med Oncol. 2020 Jul 17;12:1758835920937953. doi: 10.1177/1758835920937953. eCollection 2020. PMID 32733606
- [Background] Pan Z, Yang G, Cui J, Li W, Li Y, Gao P, Jiang T, Sun Y, Dong L, Song Y, Zhao G. A Pilot Phase 1 Study of Intrathecal Pemetrexed for Refractory Leptomeningeal Metastases From Non-small-cell Lung Cancer. Front Oncol. 2019 Aug 30;9:838. doi: 10.3389/fonc.2019.00838. eCollection 2019. PMID 31544065
- [Background] Yang JCH, Kim SW, Kim DW, Lee JS, Cho BC, Ahn JS, Lee DH, Kim TM, Goldman JW, Natale RB, Brown AP, Collins B, Chmielecki J, Vishwanathan K, Mendoza-Naranjo A, Ahn MJ. Osimertinib in Patients With Epidermal Growth Factor Receptor Mutation-Positive Non-Small-Cell Lung Cancer and Leptomeningeal Metastases: The BLOOM Study. J Clin Oncol. 2020 Feb 20;38(6):538-547. doi: 10.1200/JCO.19.00457. Epub 2019 Dec 6. PMID 31809241